# 初治成人急性髓系白血病患者中标准 "3+7" 方案与维奈克拉联合 CACAG 方案的全国多中心前瞻随机对照研究

## 知情同意书

版本号: v1.1 版本 日期: 2024 年 4 月 10 日

#### 尊敬的受试者:

我们在此邀请您参加一项临床研究:初治成人急性髓系白血病患者中标准"3+7"方案与维奈克拉联合 CACAG 方案的全国多中心前瞻随机对照研究。本知情同意书提供给您一些信息以帮助您决定是否参加此项研究。请您用一定的时间仔细阅读下面的内容,如有不清楚的问题或术语,可以与有关医生进行讨论。

您参加本项研究是完全自愿的。本研究已经得到解放军总医院第五医学中心伦理审查小组的审查和批准。

## 为什么要开展本项研究?

## 研究背景:

西达本胺、阿扎胞苷、阿克拉霉素、阿糖胞苷、重组人粒细胞集落刺激因子、维奈克 拉均是由国家食品药品监督管理局批准的药物,在我国广泛使用已经有多年历史;主要适 用于恶性血液病化疗等。目前如何进一步提高成人急性髓系白血病总体疗效,减少疾病复 发,改善总体预后是血液科医护人员面临的重点难题。

#### 研究目的:

提高急性髓系白血病患者治疗的缓解率,降低不良事件发生的概率,达到改善患者预后,延长患者生存期的目的。

#### 研究内容:

#### 1) 研究概况

本研究为多中心前瞻、随机、对照临床研究,观察 CACAG+维奈克拉方案(西达本胺+阿扎胞苷+阿克拉霉素+阿糖胞苷+重组人粒细胞集落刺激因子+维奈克拉)对初诊 AML 患者的疗效与安全性,对照组应用标准 "3+7"的 IA 方案(去甲氧柔红霉素联合阿糖胞苷)。对照组:80 例,接受经典 "3+7" IA 诱导缓解方案;试验组:80 例,接受 CACAG+维奈克拉诱导缓解方案。"随机"表示您会被随机地分配到一个治疗组中,以减少偏差。您有1/2 的机会进入对照组,1/2 的机会进入试验组,具体的分组会通过计算机程序随机确定。无论是您还是 您的医生均不能选择您接受哪种药物。这样可以保证以公正的方式对研究药物进行评估。

如果您自愿决定参加本研究,医生将检查您是否符合参加本研究的条件,询问您的健康情况和有关疾病情况,医生还将对您进行相应的体格检查,包括血、尿、便常规,肝、肾功、心电图等。如果您符合入选条件,您将随机接受试验组维奈克拉联合 CACAG 方案或者对照组 IA 方案治疗。整个试验治疗期共 1 周,每 4 周是一个治疗周期,总共 2 个疗程。

在您治疗过程中,请您按医生要求提供临床需要记录的有关信息。如果您完全自愿参加本研究,我们希望您能坚持治疗,以协助我们完成本项研究任务。如果您在任何时候因任何原因退出本研究,请与您的医生联系,并完成医生所要求回答的问题,以便能完成最后一次就诊要求的所有检查项目。如果您决定退出本试验将不会影响您与医生的关系,医生将根据您的病情和患者至上的原则对您进行其它合理治疗。

在整个研究过程中,我们将通过一系列检查和步骤来收集您对研究药物的反应和您的健康状况。

#### 2) 研究程序

本研究随访将持续3个月,在此期间,您需要来医院做一些检查、按日程进行回访,并

告诉我们您的任何变化。

- 1. 在接受试验治疗前 1 周内进行筛选期的血常规、血生化检查;
- 2. 每4周至少检查1次,可根据病情需要增加频率,包括骨髓细胞形态学分析、免疫分析等;
- 3. 适用于育龄期女性;
- 4. 在初诊时采集 5ml 骨髓样本,提取单个核细胞, -80 摄氏度冰箱保存;
- 5. 每个访视周期的窗口期为±2天。若患者治疗过程中有暂停用药,新周期开始的定义是服用新周期的试验药物。 C: 周期; W: 周; D: 天;
- 6. 结束试验治疗后 2 周内,需要返院进行结束治疗的访视;
- 7. 每 2-3 个月电话或当面随访患者的生存情况,可以通过电话随访完成。

## 其他的治疗选择

参加本研究可能改善或不能改善您的健康状况,目前的标准治疗为"3+7"的 IA 方案(去甲氧柔红霉素联合阿糖胞苷),请与您的医生协商您的决定。

## 该研究可能会带来的影响

您可能会觉得这些访视和检查会带来不便,并且需要特殊的安排。如果您有关于研究中 检查和步骤的任何疑问可以向您的研究医生咨询。

您的研究医生会告知您在研究期间哪些药物能服用,哪些药物不能服用。在服用任何新 的处方药物前请咨询您的研究医生。

如果您需要停用药物,为确保您的的安全,您需咨询研究医生怎样停用药物。

如果您是有生育能力的妇女,需要您在整个研究期间避孕,请咨询您的研究医生以确定采用的避孕方式及使用时间,研究期间某些避孕方式是不被认可的。

在整个研究期间您不能再参加其他任何有关药物或者医疗器械的临床研究。

#### 研究的风险和不良反应

您在自愿参加临床研究过程中,可能会出现一些不良反应如骨髓抑制、感染、出血、头痛、眩晕、皮疹、搔痒、胃肠道不适及过敏反应,严重时可能危及生命。如果出现,我们将予以及时、相应的治疗。如出现严重不良反应,必要时终止治疗。您在访视之间出现任何不良反应,请及时给您的研究医生打电话咨询。我们会监测研究中所有病人的任何不良反应。

#### 研究获益

参加本项研究并不会获得报酬或补偿。

#### 生物标本和医疗信息的处理和利用

本项研究将会采集受试者血液及骨髓,用于药物诱导组蛋白释放后,新填充组蛋白的表观遗传修饰特征研究、下游基因表达谱的变化特征及与组蛋白表观遗传修饰特征的融合分析,本次研究中获得的生物样本不会被二次利用。

本研究将采取匿名化处理的方式,即研究者销去除病历或标本上个人标识符的计划;受试者拥有要求对生物标本、病历、或他们认为特别敏感的病历部分(如照片、录像带或录音磁带)进行销段或匿名的权利。

研究者对获得"同意"的生物标本进行标记、保存; 医疗信息将被保存5年。

#### 您的权利和义务

您有充分的时间考虑和随时提问的权利,且是否要参加本研究的最终决定权在您。如果您决定不参加本研究,也不会影响您应该得到的其他医学关注;如果您决定参加,请您如实的告诉研究医生有关自身病史和身体状况的真实情况,告诉研究医生自己是否曾参与其他研究,或目前正参与其他研究,并请您在这份书面知情同意书上签字。签字后,您仍然可以在研究的任何阶段退出本研究。如果在研究期间发现任何新的、重要的,并且可能会影响您继续参加这一研究意愿的信息,您的研究医生或其他研究小组成员会立即通知您。您也可以随

时了解和咨询研究情况。

如果您没有遵守研究计划,或者研究医生认为您继续参加本研究不符合您的最大利益,研究医生可以让您退出研究;如果您出现了对研究药物的不良反应,或研究期间有关于研究药物的新的安全性的信息出现,研究医生或申办者可能会在未征得您同意的情况下终止您参与本项研究。如果您因为某些原因从研究中退出,您可能被询问有关您使用研究药物的情况。如果研究医生认为需要,您也可能被要求进行计划外的体格检查和实验室检查,研究医生将会和您讨论退出研究后的医疗事宜。

### 报酬或补偿

参加本项研究并不会获得报酬或补偿。

#### 研究所致损害的处理措施

西达本胺、阿扎胞苷、阿克拉霉素、阿糖胞苷、重组人粒细胞集落刺激因子、维奈克拉 均是由国家食品药品监督管理局批准的药物,在我国广泛使用已经有多年历史。如果您的健康确因参加这项研究而发生与研究相关的损害,请立即通知研究医生,研究医生将负责对您 采取适当的治疗措施。

即使您已经签署这份知情同意书,您仍然保留您所有的合法权利。如您的权益受到侵犯,您可以联系中国人民解放军总医院第五医学中心伦理审查小组,电话:010-66947798。

#### 保密性

如果您决定参加本项研究,您参加研究及在研究中的个人资料均会保密。负责研究的医生及其他研究人员将使用您的医疗信息进行研究。您的档案仅供研究人员查阅。研究中会用编号来标识您的研究信息和实验室检查标本。您的身份不会被识别,只有研究医生和研究小组成员可查询编号。

为确保研究按照规定进行,必要时,政府管理部门或伦理审查委员会的成员按规定可以 在研究单位查阅您的个人资料,此过程中不会泄露您的任何信息。任何有关本项研究结果的 公开报告均不会披露您的个人身份。

我们将遵循有关法律和规定,确保您个人医疗资料的隐私得到充分保护。

#### 自愿参加

参加本研究是完全自愿的,您可以拒绝参加研究,或者研究过程中的任何时候选择退出研究,不需任何理由。该决定不会影响您未来的治疗。如果您决定退出本研究,请提前通知您的研究医生。为了保障您的安全,您可能被要求进行相关检查,这对保护您的健康是有利的。

#### 研究中如何获得帮助:

您可随时了解与本研究有关的信息资料和研究进展,如果您有与本研究有关的问题,请联系 \_\_\_\_\_(电话号码)与\_\_\_\_\_(研究者或有关人员姓名)联系。如果您在研究过程需要了解关于本项研究受试者权益方面的问题您可以联系中国人民解放军总医院第五医学中心伦理审查小组,电话:010-66947798。

## 知情同意签字页

#### 受试者声明:

我在充分了解该项研究的知情同意书的全部内容以及参加本研究可能带来的风险和受益后,自愿参加本试验,并做出以下申明:

- 1. 我已阅读了上述知情同意书中的内容并理解本研究的性质、目的及该项研究可能出现的不良反应等信息,我的问题已经得到满意的答复。
- 2. 我将遵守知情同意书中要求,并与研究人员充分合作,如实、客观地向研究人员提供参加本研究前、研究期间和各随访期的健康状况及相关情况。
- 3. 我明白我可以随时退出研究,而此后的治疗并不会因此受到任何不利影响。我理解研究者有权根据我的情况随时终止研究。
- 4. 我知晓我会收到一份签署过的知情同意书。
- 5. 我已得知参与本研究的医生、相关主管部门的负责人以及中国人民解放军总医院第五医学中心伦理审查小组均有权审阅研究记录和病例资料,我同意上述方面的人员直接得到我的研究记录,并了解上述 信息将得到保密处理。
- 6. 经过充分考虑后,我自愿参加本临床研究。

| 文试有金名:<br> | 口别: |
|----------------------------------------------------------------|-----|
| 联系电话: | |
| 监护人者签名: | |
| 联系电话: | - |
| 公平见证人: | 日期: |
| 联系电话: | _ |
| 研究者声明: | |
| 我确认已向患者解释了本研究的详细情况,特别是参加本研究可能产生的风险和受益,并给受试者一份双方签署过姓名和日期的知情同意书。 | |
| 研究者签名: | 日期: |
| 研究者联系由话: | |